CLINICAL TRIAL: NCT02403921
Title: Association Between Cortisol, Cortisone, Cotinine, Nicotine, Caffeine, Melatonin Levels in Hair, Serum, Urine, Saliva and Chronic Stress
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201412205RINA
Record Dates: First submitted 2015-03-26; First posted 2015-03-31 (Estimated); Last update posted 2015-03-31 (Estimated); Status verified 2015-03

CONDITIONS: Hydrocortisone
Keywords: biomarker

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators aim to investigate the association between hair, serum, urine and saliva to measure cortisol, cortisone, cotinine, nicotine, melatonin and caffeine.

ELIGIBILITY:
Inclusion Criteria:

* adult volunteer

Exclusion Criteria:

* students of the study host
* people who have steroid or melatonin medicine

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: adult volunteer
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2015-03; Primary Completion 2016-01 (Estimated); Study Completion 2016-01 (Estimated)

PRIMARY OUTCOMES:
Chinese Health Questionnaire (CHQ) | 5 minutes
Hospital Anxiety and Depression Scale (HADS) | 5 minutes
Pittsburgh Sleep Quality Index (PSQI) | 5 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Pau-Chung CHEN, Principal Investigator — National Taiwan University
Locations (1):
- National Taiwan University Hospital, Test1, Test2, Taiwan